CLINICAL TRIAL: NCT01926171
Title: A Single Center, Open Label, Multicenter Study to Determine the Safety and Efficacy of Icotinib in Combination With Whole Brain Radiation Therapy For NSCLC Patients With Brain Metastases
Brief Title: Icotinib With Whole Brain Radiation Therapy in NSCLC Patients With Brain Metastases
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IV-49
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib plus WBRT (Experimental): Standard whole brain radiotherapy is given with 4000cGY/20 times, plus concurrent icotinib, which was administered orally three times per day.
  Interventions: Drug: Icotinib plus WBRT

INTERVENTIONS:
Drug: Icotinib plus WBRT — Standard whole brain radiotherapy is given with 4000cGY/20 times, plus icotinib, which was administered orally three times per day.
  Other Names: Commana; BPI-2009

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of icotinib in combination with whole brain radiotherapy for NSCLC patients with brain metastases. The primary endpoint is objective response rate of intracranial lesions.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is one of the malignant tumors with the highest incidence of brain metastases. Patients with multiple brain metastasis showed poor prognosis and displayed an untreated median survival of only 3-6 months, and most patients died due to the progression of brain metastases. This study is designed to evaluate the safety and efficacy of icotinib combined with whole brain radiotherapy for NSCLC patients with brain metastases. The primary endpoint is intracranial objective response rate .

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of non-small-cell lung cancer (NSCLC).
* Diagnosis of non-systematic brain metastases on a Gadolinium-enhanced MRI. More than 2 sites of intracranial metastases, or the longest diameter of the intracranial lesion is more than 3cm.
* No other metastases except for brain metastases.

Exclusion Criteria:

* Previous usage of EGFR-TKI or antibody to EGFR: gefitinib, erlotinib, herceptin, erbitux.
* CSF or MRI findings consistent with metastases of spinal cord, meninges or meningeal.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate of intracranial lesions | 8 weeks
  Number of participants with an objective response. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to RECIST, confirmed at least 28 days following the date of the initial response.

SECONDARY OUTCOMES:
Objective response rate of extracranial lesions | 8 weeks
  Number of participants with an objective response of extracranial lesions. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to RECIST, confirmed at least 28 days following the date of the initial response.
Progression-free survival of intracranial lesions | 3-6 months
  All cause progress or mortality
Safety and tolerability | 6-12 months
  All cause adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhu, MD, Principal Investigator — Baotou Central Hospital
Locations (1):
- Baotou Central Hospital, Baotou, Inner Mongolia, China